CLINICAL TRIAL: NCT00004785
Title: Phase III Randomized, Double-Blind Study of Dexamethasone Vs Dexamethasone/Methylprednisolone Vs Placebo for Bronchopulmonary Dysplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Iowa (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11874; UIHC-69501
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; cardiovascular and respiratory diseases; neonatal disorders; rare disease
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Respiratory Tract Diseases; Infant, Newborn, Diseases; Rare Diseases | interventions — Dexamethasone; Methylprednisolone

INTERVENTIONS:
Drug: dexamethasone
Drug: methylprednisolone

SUMMARY:
OBJECTIVES: I. Compare the efficacy of dexamethasone (DM) vs. DM/methylprednisolone treatment vs. placebo, initiated within the first month of life, on long-term pulmonary and developmental outcomes in premature infants with evolving bronchopulmonary dysplasia.

II. Compare the toxicities of these treatments. III. Assess treatment effects on adrenal function.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are randomly assigned to 1 of 3 treatment groups. The first group receives intravenous dexamethasone tapered over 42 days.

The second group receives daily intravenous dexamethasone for 6 days, then intravenous methylprednisolone (MePRDL) tapered over the next 34 days, beginning on day 8. A placebo is given on "off" MePRDL days.

The third group receives an intravenous placebo for 42 days, with a tapering schedule beginning day 35.

All patients may receive 6 days of dexamethasone rescue therapy beginning day 15 and/or 30, as clinically indicated. Study drugs are suspended during rescue therapy.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Premature infants with evolving bronchopulmonary dysplasia on chest x-ray Requirement for mechanical ventilation Fraction of inspired oxygen greater than 0.30 Ventilator at least 15 cycles/minute No signs of weaning within 72 hours prior to entry No serious congenital anomaly --Prior/Concurrent Therapy-- No prior postnatal corticosteroids --Patient Characteristics-- Cardiovascular: No congenital heart disease Other: Birth weight no greater than 1500 g Gestational age no greater than 30 weeks No contraindication to corticosteroids, e.g., culture-proven bacterial sepsis

Ages: 0 Years to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54
Dates: Start 1995-11

CONTACTS AND LOCATIONS:
Overall Officials: Richard C. Ahrens, Study Chair — University of Iowa